CLINICAL TRIAL: NCT03085459
Title: The Effect of Nursing Staff on Empiric Antibiotic Treatment Within the First Hour in Patients With Septic Shock: A Retrospective Study
Brief Title: Effects of Nursing Staff on Empiric Antibiotic in Septic Shock
Status: Completed | Type: Observational
Sponsor: Chun Pan (Other)
Responsible Party: Sponsor-Investigator, Chun Pan, Principal Investigator, Southeast University, China
Organization: Southeast University, China (Other)
Other Study IDs: Nurse: empiric antibiotic
Record Dates: First submitted 2017-01-31; First posted 2017-03-21 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Septic Shock; Compliance; Antibiotic; Nursing Caries
MeSH Terms: conditions — Shock, Septic; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Nurse level N0: who got college degree or above, nurse qualification certificate and working time less than one year
  Interventions: Behavioral: work Time
- Nurse level N1: who got nurse qualification certificate and working time between 1~3 years
  Interventions: Behavioral: work Time
- Nurse level N2: who got nurse qualification certificate and working time between 3~5 years
  Interventions: Behavioral: work Time
- Nurse level N3: who got nurse qualification certificate and working time more than 5 years
  Interventions: Behavioral: work Time

INTERVENTIONS:
Behavioral: work Time — nurse got qualification certificate and the working time

SUMMARY:
A retrospective, observational study was performed about the patients with septic shock who admitted into intensive care unit (ICU) from January 1, 2015 to February 29, 2016. The number of patients who received empiric antibiotic treatment within first hour after septic shock diagnosis were collected. Detailed information about clinical ladder for nursing stuff and nursing shift were collected . Clinical ladder for nursing stuff is a new definition based on education background and work experience and nurses stuff are classified into four levels. N0 was defined who got college degree or above, nurse qualification certificate and working time less than one year. N1 an N2 were defined as who got nurse qualification certificate and working time between 1~3 years and more than three years, respectively. N3 was defined who was nurse-in-charge qualification or got nurse practitioner qualification for more than five years. Compliance of empiric antibiotic treatment within first hour and evaluate the effect of nursing stuff on the compliance were calculated.

ELIGIBILITY:
Inclusion Criteria:

* age>18 years old
* sepsis

Exclusion Criteria:

* pregnancy
* >80 years old.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients whose age of 18 years or older admitted to the ICU with septic shock from between January 01, 2015 to February 29, 2016
Sampling Method: Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2015-01-12 (Actual); Primary Completion 2016-02-29 (Actual); Study Completion 2016-02-29 (Actual)

PRIMARY OUTCOMES:
compliance of empiric antibiotic treatment within first hour | 1 hour
  compliance of empiric antibiotic treatment within first hour
evaluate the effect of nursing stuff on the compliance | 1 hour
  evaluate the effect of nursing stuff on the compliance

IPD SHARING:
Plan to Share IPD: No